CLINICAL TRIAL: NCT03005392
Title: Effects of a Physical Exercise Program in Patients With Diagnosis of Acute Lymphoblastic Leukemia
Brief Title: Home-exercise Program for Children and Adolescent Survivors of Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-EJE-2013-150
Record Dates: First submitted 2016-12-13; First posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Cancer; Physical therapy; Cardiorespiratory fitness
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Evaluate physical fitness (Experimental): An exercise program will be designed over 16 weeks with 55 sessions, moderately increasing the volume and intensity of the load every 4 weeks. The program will consist of strength exercises, flexibility and aerobic endurance, which will be explained in videos and are going to be available in an online platform
  Interventions: Other: exercise
- Evaluate Cardiological changes (Experimental): An exercise program will be designed over 16 weeks with 55 sessions, moderately increasing the volume and intensity of the load every 4 weeks. The program will consist of strength exercises, flexibility and aerobic endurance, which will be explained in videos and are going to be available in an online platform
  Interventions: Other: exercise
- Evaluate activity physical (Experimental): An exercise program will be designed over 16 weeks with 55 sessions, moderately increasing the volume and intensity of the load every 4 weeks. The program will consist of strength exercises, flexibility and aerobic endurance, which will be explained in videos and are going to be available in an online platform
  Interventions: Other: exercise
- control grup (No Intervention): The control group will be recommended to maintain a level of physical activity they would routinely and habitually have during the 4 months that the study will last.

INTERVENTIONS:
Other: exercise — An exercise program will be designed over 16 weeks with 55 sessions, moderately increasing the volume and intensity of the load every 4 weeks. The program will consist of strength exercises, flexibility and aerobic endurance, which will be explained in videos and are going to be available in an online platform.
  The physiotherapist will contact the patient and/or tutor weekly so as to answer and doubts they may have with respect to the exercise program and to further supervise their compliance (group with intervention).
  Arms: Evaluate Cardiological changes; Evaluate activity physical; Evaluate physical fitness

SUMMARY:
* Exercise programs in children and teenagers with Acute Lymphoblastic Leukemia (ALL) strengthens their physical fitness.
* Exercising improves muscular and functional mobility fitness after finalizing chemotherapy in children and teenagers diagnosed with ALL.
* Assess cardiological changes

DETAILED DESCRIPTION:
Children and adolescents survivors of ALL will be randomly assigned to the intervention group and to the control group. A home-exercise program will be designed for 16 weeks with 55 sessions, combining aerobic, strength and flexibility exercises of light and moderate intensity. The following tests will be performed to evaluate the effects of the intervention program: Echocardiography, Tape treadmill test using a ramp protocol to assess cardiorespiratory fitness, hand grip test to assess muscular grip strength, Timed Up test And Go Test (TUG) and Timed Up and Down Stairs Test (TUDS) to assess functional mobility, the sit and reach test to assess flexibility and a questionnaire to assess levels of physical activity. The control group will perform their usual physical activity

ELIGIBILITY:
Inclusion Criteria:

* The study included of children and adolescents between 7 and 18 years old that were at time in complete remission for a minimum of one year of their neoplastic disease and had finalized their chemotherapy treatments by the time they began the physical exercise program.

Exclusion Criteria:

* Patients with structural cardiac anomalies, congenital cardiopathies, those in recurrence of their neoplastic diseases, signs of clinical or subclinical cardiac insufficiency and an echocardiography with alterations in systolic and/or diastolic function.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory exercise test | 1 year
  For this test a treadmill was used utilizing a sloped ramp protocol

SECONDARY OUTCOMES:
Echocardiography | 1 year
  Index of the lateral mitral annulus level (isovolumetric contraction time
  + Isovolumetric relaxation time / ejection time), measured by Echocardiography. Index of TEI at the level of the septal mitral ring (isovolumetric contraction time + Isovolumetric relaxation time / ejection time), measured by means of Echocardiography. TEI index at the level of the tricuspid ring (isovolumetric contraction time + Isovolumetric relaxation time / ejection time), measured by means of Echocardiography.
Functional mobility | 1 year
  For this variable the Time Up and Go Test (TUG) was used
Functional mobility | 1 year
  For this variable the Time Up and Down Stairs Test (TUDS) was used
Strength | 1 year
  To measure this variable, the hand grip test was utilized
Flexibility | 1 year
  For this variable the sit-and-reach (SR) test was used, that of which allowed evaluation of the hamstring muscle extensibility
Level of physical activity | 1 year
  This variable was measured utilizing the family of the international questionnaire of physical activity (IPAQ). For children between the ages of 8-12 the Physical Activity Questionnaire for Children (PAQ-C) version was used, and for adolescents between the ages of 13-18 the PAQ-A form was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Claudia Delgado, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] R. Peris-Bonet, D. Salmerón, M. A. Martínez-Beneito, J. Galceran, R. Marcos Gragera, S. Felipe, V. González & J. Sanchez de Toledo Codina. Childhood cancer incidence and survival in Spain. Annals of Oncology 2010: 21 arner JT.; Bell W.; Webb DK.; Gregory JW. Daily energy expenditure and physical activity in survivors of childhood malignancy. Pediatr Res 43. 1998, 607-613 Lucia A.; Earnest C.; Perez M. Cancer-related fatigue: can exercise physiology assist oncologists?. Lancet Oncol 4. 2003, 616-625 San Juan AF.; Fleck SJ.; Chamorro C.; Maté-Muñoz JL.; Garcia-Castro J.; Ramirez M.; Madero L.; Lucia A. Early-phase adaptations to intra-hospital training in strength and functional mobility of children with Leucemia.J Strength Cond Res. 2006